CLINICAL TRIAL: NCT05093504
Title: Safe & Timely Antithrombotic Removal-Direct Oral Anticoagulants (STAR-D): Prospective, Multicenter, Double-blind, Randomized Study of Apixaban & Rivaroxaban Removal to Reduce Risk of Serious Bleeding in Urgent Cardiac Surgery Patients
Brief Title: Safe and Timely Antithrombotic Removal - Direct Oral Anticoagulants Apixaban & Rivaroxaban (STAR-D)
Acronym: STAR-D
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision for business reasons.
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-02
Record Dates: First submitted 2021-10-01; First posted 2021-10-26 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hemorrhage, Surgical; Hemorrhage Postoperative; Blood Loss, Surgical; Blood Loss, Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control (Sham Comparator): Standard of care with Sham set-up
  Interventions: Device: Sham comparator
- DrugSorb-ATR Intervention (Experimental): Standard of care + DrugSorb-ATR system
  Interventions: Device: DrugSorb-ATR system

INTERVENTIONS:
Device: Sham comparator — Sham comparator in similar position to the investigational device, but NOT integrated into the cardiopulmonary bypass (CPB) circuit
  Arms: Control
Device: DrugSorb-ATR system — Sorbent hemoperfusion system integrated into the cardiopulmonary bypass (CPB) circuit
  Other Names: Sorbent hemoperfusion system
  Arms: DrugSorb-ATR Intervention

SUMMARY:
Prospective, Multicenter, Double-blind, Randomized, Study to Evaluate DrugSorb-ATR Removal of Apixaban and Rivaroxaban to Reduce Likelihood of Serious Bleeding in Patients Undergoing Urgent Cardiothoracic Surgery

DETAILED DESCRIPTION:
The Safe and Timely Antithrombotic Removal - Direct Oral Anticoagulants (DOACs) Apixaban & Rivaroxaban (STAR-D) study is a prospective, multicenter, double-blind, randomized study that evaluated the DrugSorb™-Antithrombotic Removal (ATR) device for removal of apixaban and rivaroxaban to reduce the likelihood of serious bleeding in patients undergoing urgent cardiothoracic surgery. The objectives were

* To demonstrate reductions in surgical and early post-surgical bleeding with the intraoperative use of DrugSorb-ATR in patients undergoing cardiothoracic surgery ≤36hrs since last apixaban or rivaroxaban dose.
* To demonstrate reductions in apixaban or rivaroxaban blood levels (Δ[DOAC]) with the intraoperative use of DrugSorb-ATR.
* To establish the safety of the intraoperative use of DrugSorb-ATR in the intended population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older, with documented full, written informed consent
2. Requiring cardiothoracic (CT) surgery with cardiopulmonary bypass (CPB) within 36 hours from last dose of either apixaban or rivaroxaban (*note that patients must be taking apixaban or rivaroxaban for one of the following indications: a) reduction of stroke/systemic embolism in nonvalvular atrial fibrillation, or b) initial or extended treatment of venous thromboembolism)

Exclusion Criteria:

1. >48hrs between last apixaban or rivaroxaban dose and start of CT surgery
2. Patients on low dose apixaban or rivaroxaban for prophylactic indications
3. Heart-lung transplant procedures
4. Procedures for ventricular assist device (i.e., implant or revision of left ventricular assist device [LVAD] or right ventricular assist device [RVAD])
5. Any of the below conditions that pose a known risk for increased bleeding

   1. Heparin induced thrombocytopenia
   2. Preoperative platelet count <50,000u/L
   3. Hemophilia
   4. International normalized ratio (INR) greater than or equal to 1.8
6. Prohibited concomitant antithrombotic medications as defined in the study protocol
7. Acute sickle cell crisis
8. Known allergy to device components
9. Active (untreated) systemic infection
10. History of major organ transplantation and those currently receiving immunosuppressive medication or who are profoundly immune suppressed
11. Women with positive pregnancy test during current admission or who are breast-feeding
12. Life expectancy <30 days
13. Inability to comply with requirements of the study protocol
14. Treatment with investigational drug or device within 30 days of current surgery
15. Previous enrollment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mack, MD, Principal Investigator — Baylor Scott & White The Heart Hospital; C. M Gibson, MD, Principal Investigator — Beth Israel Deaconess Medical Center, The Baim Institute, and Harvard Medical School
Locations (27):
- United States (27):
  - University of California, Davis Medical Center, Sacramento, California
  - University of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Baptist Hospital of Miami and its Miami Cardiac and Vascular Institute, Miami, Florida
  - Advent Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital Midtown/Emory School of Medicine, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Lutheran Medical Group, Fort Wayne, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi, Jackson, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Bryan Medical Center, Lincoln, Nebraska
  - Virtua Health, Marlton, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Bethesda North Hospital, TriHealth, Inc, Cincinnati, Ohio
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott & White The Heart Hospital, Plano, Texas
  - VCU Medical Center, Richmond, Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tripathi R, Morales J, Lee V, Gibson CM, Mack MJ, Schneider DJ, Douketis J, Sellke FW, Ohman ME, Thourani VH, Storey RF, Deliargyris EN. Antithrombotic drug removal from whole blood using Haemoadsorption with a porous polymer bead sorbent. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 2;8(8):847-856. doi: 10.1093/ehjcvp/pvac036. PMID 35657375

RESULTS

PARTICIPANT FLOW:
Groups:
- DrugSorb-ATR Intervention: Standard of care + DrugSorb-Antithrombotic Remove (ATR) system
  DrugSorb-ATR system: Sorbent hemoperfusion system integrated into the cardiopulmonary bypass (CPB) circuit
Period: Overall Study
Arm/Group | Control | DrugSorb-ATR Intervention
Started | 5 | 4
Completed | 5 | 3
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | DrugSorb-ATR Intervention | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (14.7) | 68.5 (12.2) | 65.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Hypertension [Count of Participants; unit: Participants] | 5 | 2 | 7
Heart failure [Count of Participants; unit: Participants] | 1 | 1 | 2
Coronary artery disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Subjects with apixaban [Count of Participants; unit: Participants] | 4 | 2 | 6
Subjects with rivaroxaban [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Perioperative Bleeding
Description: Incidence of clinically significant perioperative bleeding events, as evaluated by a ranked composite endpoint
Time Frame: Through the first 48 hours post-operation
Population: The trial was terminated before the outcome measure data were cleaned and adjudicated. All bleeding outcomes data were to be adjudicated by a Clinical Events Committee, which was not convened because the trial was terminated. Therefore, no bleeding outcomes were available.
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Direct Oral Anticoagulant (DOAC) Drug Removal: Apixaban and Rivaroxaban
Description: Percent change in blood apixaban or rivaroxaban levels from pre coronary bypass (CPB), that is, start of device use to 30 min post CPB
Time Frame: Through 30 minutes post-CPB
Population: Because of the premature discontinuation of the study, this is the only outcome measure collected and analyzed. The change in drug levels was analyzed for both rivaroxaban and apixaban together (not separately), again due to the low number of enrolled subjects.
Measure: Mean (Standard Deviation); unit: percent change in drug levels
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 5 | 4
percent change in drug levels | 27.95 (8.6) | 62.21 (8.9)
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Chest Tube Drainage
Description: Drainage volume from all chest and mediastinal tubes
Time Frame: Through 24 hours post-operation
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Platelet Transfusions (Volume)
Description: Total platelet transfusions (mL) during hospitalization
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Platelet Transfusions (Units)
Description: Total platelet transfusions (units) during hospitalization
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Packed Red Blood Cell (PRBC) Transfusions (Volume)
Description: Total PRBC transfusions (mL) during hospitalization
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: PRBC Transfusions (Units)
Description: Total PRBC transfusions (units) during hospitalization
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Incidence of Moderate, Severe, and Massive Perioperative Bleeding Events
Description: Perioperative bleeding events classified according to the Universal Definition of Perioperative Bleeding, and analyzed by class (Class 0, 1, 2, 3, 4)
Time Frame: Through the first day post-operation
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Surgical Re-exploration for Bleeding
Description: All surgical re-explorations for excessive bleeding, as adjudicated by an independent Clinical Events Committee
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Population: as for outcome 1
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Fatal Perioperative Bleeding
Description: Deaths directly attributable to procedure-related bleeding.
Time Frame: Through to discharge from index hospitalization, on average 1-2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study duration, that is, within 30 days post-operation
Arm/Group | Control | DrugSorb-ATR Intervention
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/4
Other Adverse Events (participants affected / at risk) | 2/5 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=5) | DrugSorb-ATR Intervention (N=4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemi (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=5) | DrugSorb-ATR Intervention (N=4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Cortisol decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Not reported as serious adverse event (SAE)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) — Not reported as SAE
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) — Not reported as serious adverse event

LIMITATIONS AND CAVEATS:
The study was terminated early for business reasons, due to low enrollment. Outcome data was not cleaned, nor adjudicated. The only outcome available to analyze was the percent change in drug levels for both direct oral anticoagulants or DOACs rivaroxaban and apixaban together--there were not enough subjects to analyze DOAC levels separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05093504/Prot_SAP_001.pdf